CLINICAL TRIAL: NCT05345665
Title: Comparison of Three Methods of Anesthesia to Achieve a Nerve Block Anesthesia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, FAHA, Head of Department, Astes
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: DAED
Record Dates: First submitted 2022-03-26; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Echography (Other): For the neuronal blockade of the patient, anesthesiologists used an echography.
  Interventions: Other: Echography; Other: Echography and neurostimulation; Other: Echography, neurostimulation and active mobilization
- Neurostimulation (Other): For the neuronal blockade of the patient, anesthesiologists used neurostimulation.
  Interventions: Other: Echography and neurostimulation; Other: Echography, neurostimulation and active mobilization
- Active mobilization (Other): For the neuronal blockade of the patient, anesthesiologists used active mobilization.
  Interventions: Other: Echography, neurostimulation and active mobilization

INTERVENTIONS:
Other: Echography — Neuronal blockade anesthesia for elective surgery of the hand was performed with an only echography.
  Arms: Echography
Other: Echography and neurostimulation — Neuronal blockade anesthesia for elective surgery of the hand was performed with both echography and neurostimulation.
  Arms: Echography; Neurostimulation
Other: Echography, neurostimulation and active mobilization — Neuronal blockade anesthesia for elective surgery of the hand was performed with echography, neurostimulation, and active mobilization.

SUMMARY:
Evaluation of three methods for the realization of a neuronal blockade.

DETAILED DESCRIPTION:
Evaluation of three methods during the realization of a neuronal blockade. The three stimulations were: 1) echography, 2) echography and neurostimulation, and 3) echography, neurostimulation, and active mobilization by the patient.

ELIGIBILITY:
Inclusion Criteria:

* 216 consecutive adult patients scheduled for an elective hand surgery

Exclusion Criteria:

* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Time | Measurements was performed during 20 minutes after the completion of the neuronal blockade.
  Time to obtain a complete neuronal blockade of the hand

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Deflandre, MD, PhD, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc Bouge, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No